CLINICAL TRIAL: NCT06609694
Title: Comparison of a Demand Oxygen Delivery to Continuous Flow for Administration of Oxygen During Sleep
Brief Title: Comparison of a Demand Oxygen Delivery
Acronym: DOSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2022-0821; R61HL165366 (NIH)
Record Dates: First submitted 2023-01-06; First posted 2024-09-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Apnea
Keywords: Sleep Apnea; Down Syndrome; Continuous Positive Airway Pressure (CPAP)
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Down Syndrome

STUDY DESIGN:
Intervention Model Description: The aim of this study is to examine whether clinically important indices during sleep are comparable between oxygen delivery by portable and by continuous flow. This aim will be accomplished by a randomized crossover study design.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Inogen portable oxygen concentrator unit versus continuous flow (Pilot Study) (Experimental): The aim of this pilot study is to examine whether clinically important indices during sleep are comparable between oxygen delivery by portable and by continuous flow.
  Interventions: Device: Portable oxygen concentrator Inogen G5 model
- Reducing the frequency of obstructive apnea (Main study) (Experimental): The arm of the main study is still under development
  Interventions: Device: Portable oxygen concentrator Inogen G5 model

INTERVENTIONS:
Device: Portable oxygen concentrator Inogen G5 model — The concentrator weighs 4.7 lbs. and has a battery life of 13 hours. It has 6 settings with 1 providing the lowest pulse flow and 6 provides the highest flow. The setting will be increased every 30 minutes by 1 when oxygen nadir is lower than 94% and or obstructive index is ≥ 5 /hour.

SUMMARY:
Conducting a randomized control trial of oxygen in children with Down syndrome to treat moderate to severe obstructive sleep apnea.

The aim of the study is to conduct a comparison between the 2 methods of oxygen delivery during sleep in 15 children from Cincinnati Children's Hospital and Children's Hospital of Los Angeles. 2 polysomnographies will be performed, one with continuous flow and the second with pulse flow.

DETAILED DESCRIPTION:
Cincinnati Children's Hospital received NIH funding to conduct a randomized control trial of oxygen in children with Down syndrome to treat moderate to severe obstructive sleep apnea. Oxygen may be delivered through continuous flow for the duration of the respiratory cycle or pulse flow during inspiration only. Pulse flow oxygen concentrators have been used clinically in adults. However, there is limited experience with this technology in children. The advantages of pulse flow oxygen concentrator are its portability and its ability in providing compliance data.

This is a pilot research study to compare the 2 methods of oxygen delivery during sleep in 15 children from Cincinnati Children's Hospital and Children's Hospital of Los Angeles. 2 polysomnographies will be performed, one with continuous flow and the second with pulse flow. The pilot study is conducted in preparation for a larger project which will include 7 sites aiming at determining the effect of oxygen treatment on the frequency of obstructive apnea, neurocognitive and cardiac outcomes. A separate Institutional Review Board (IRB) protocol of the larger study will be submitted later once approved by the NIH Data and Safety Monitoring Board.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5-17 years with or without Down Syndrome (DS).
2. Children with obstructive sleep apnea (OSA) and obstructive apnea hypopnea index (OAHI) 5-40 / hour: The rationale for selecting this range of OAHI is that a large number of children with DS with this range of OSA severity are untreated for months to years. It is important to understand the response to oxygen across the spectrum of disease severity. Notably, children with severe disease are left with few options (e.g., tracheostomy).
3. Absence of clinically significant hypoxia defined as oxygen saturation < 88% for 5 minutes or episodic desaturation to 60% as these levels would otherwise identify children eligible to routinely receive oxygen.

Exclusion Criteria:

1. Current CPAP use with documented compliance (> 4 hrs/ night; > 70% of nights).
2. Oxygen saturation < 90% at rest during wakefulness
3. Chronic daytime or nighttime use of supplemental oxygen.
4. Unable to participate in a Polysomnogram (PSG).
5. Enrolled or planning to enroll in another study that may conflict with protocol requirements or confound results in this trial.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Drop in Apnea Hypopnea Index (0-4 /night) by 50 % or < 5 /hour | 6 months
  Percent of children with a drop in Apnea Hypopnea Index (AHI) by 50% or < 5 /hour

SECONDARY OUTCOMES:
Value of Oxygen Saturation (SpO2) | 6 months
  The total value of how much oxygen saturation happens while sleeping will be measured at baseline and 6 month visit.
Percentage of Oxygen Saturation (SpO2) and number of times it goes below 90% | 6 months
  At the baseline and 6 month visit will measure the number of times that SpO2 falls below 90% will sleeping.
Pulse Rate during sleep | 6 months
  Mean pulse rate during the total sleep time (beats per min) as well as the maximum pulse rate will be captured during sleep.
Frequency of apnea happening during sleep | 6 months
  The total number of apnea events occurring per hour will be measured during sleep
Total hours of Sleep Time | 6 months
  Total sleep time will be confirmed by an electroencephalogram (h)

CONTACTS AND LOCATIONS:
Overall Officials: Raouf Amin, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
The primary goal of this study is to assess feasibility of using pulse oxygen flow in children with Down syndrome and obstructive sleep apnea population. Preliminary data on the response rates from the two concentrators will be obtained and a confidence interval for the difference in response rate will be obtained. Data that is obtained from the devices will be shared with Inogen. Data will be deidentified prior to sending.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year
Access Criteria: Pending

REFERENCES:
- [Background] Liu JP, Hsueh HM, Hsieh E, Chen JJ. Tests for equivalence or non-inferiority for paired binary data. Stat Med. 2002 Jan 30;21(2):231-45. doi: 10.1002/sim.1012. PMID 11782062
- [Result] Chamseddin BH, Johnson RF, Mitchell RB. Obstructive Sleep Apnea in Children with Down Syndrome: Demographic, Clinical, and Polysomnographic Features. Otolaryngol Head Neck Surg. 2019 Jan;160(1):150-157. doi: 10.1177/0194599818797308. Epub 2018 Aug 28. PMID 30149781
- [Result] Lee CF, Lee CH, Hsueh WY, Lin MT, Kang KT. Prevalence of Obstructive Sleep Apnea in Children With Down Syndrome: A Meta-Analysis. J Clin Sleep Med. 2018 May 15;14(5):867-875. doi: 10.5664/jcsm.7126. PMID 29734982
- [Result] Waters KA, Castro C, Chawla J. The spectrum of obstructive sleep apnea in infants and children with Down Syndrome. Int J Pediatr Otorhinolaryngol. 2020 Feb;129:109763. doi: 10.1016/j.ijporl.2019.109763. Epub 2019 Nov 1. PMID 31704574
- [Result] Nerfeldt P, Sundelin A. Obstructive sleep apnea in children with down syndrome - Prevalence and evaluation of surgical treatment. Int J Pediatr Otorhinolaryngol. 2020 Jun;133:109968. doi: 10.1016/j.ijporl.2020.109968. Epub 2020 Feb 26. PMID 32126418
- [Result] Shete MM, Stocks RM, Sebelik ME, Schoumacher RA. Effects of adeno-tonsillectomy on polysomnography patterns in Down syndrome children with obstructive sleep apnea: a comparative study with children without Down syndrome. Int J Pediatr Otorhinolaryngol. 2010 Mar;74(3):241-4. doi: 10.1016/j.ijporl.2009.11.006. Epub 2010 Jan 25. PMID 20097432
- [Result] MacDonagh L, Farrell L, O'Reilly R, McNally P, Javadpour S, Cox DW. Efficacy and adherence of noninvasive ventilation treatment in children with Down syndrome. Pediatr Pulmonol. 2021 Jun;56(6):1704-1715. doi: 10.1002/ppul.25308. Epub 2021 Mar 17. PMID 33730448
- [Result] Trucco F, Chatwin M, Semple T, Rosenthal M, Bush A, Tan HL. Sleep disordered breathing and ventilatory support in children with Down syndrome. Pediatr Pulmonol. 2018 Oct;53(10):1414-1421. doi: 10.1002/ppul.24122. Epub 2018 Jul 10. PMID 29992744
- [Result] Amaddeo A, Khirani S, Griffon L, Teng T, Lanzeray A, Fauroux B. Non-invasive Ventilation and CPAP Failure in Children and Indications for Invasive Ventilation. Front Pediatr. 2020 Oct 26;8:544921. doi: 10.3389/fped.2020.544921. eCollection 2020. PMID 33194886
- [Result] Dudoignon B, Amaddeo A, Frapin A, Thierry B, de Sanctis L, Arroyo JO, Khirani S, Fauroux B. Obstructive sleep apnea in Down syndrome: Benefits of surgery and noninvasive respiratory support. Am J Med Genet A. 2017 Aug;173(8):2074-2080. doi: 10.1002/ajmg.a.38283. Epub 2017 May 24. PMID 28544488